CLINICAL TRIAL: NCT01210573
Title: Prospective Observation of Exercise Parameters in Advanced Heart Failure
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: Shape Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1002M77542
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Advanced Heart Failure
Keywords: Heart Failure; Heart-Assist Devices; Left Ventricular Assist Device
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy Devices

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Device adjustment: Advanced or suspected advanced heart failure. Most are anticipated to have severely depressed ejection fraction (<30% and typically <20%), but patients with preserved ejection fraction and either hypertrophy or restrictive cardiomyopathy will also be eligible. Patients pulmonary hypertension, on any therapy (other than diuretics alone), are also felt to be at high risk of developing right heart failure and may also be included. Patients who have already undergone LVAD or cardiac transplant are also considered to have advanced heart failure and are eligible to participate, regardless of the severity of their symptoms at the time of enrollment.
  Interventions: Device: adjustment of LVAD or pacemaker

INTERVENTIONS:
Device: adjustment of LVAD or pacemaker — For patients without a device: Patients start at rest for 2 minutes and will wear a face mask and breathing parameters are recorded using the SHAPE-HF system (SHAPE Medical St. Paul, MN) that measures respiratory airflow and the constituent respiratory gases, oxygen and carbon dioxide.
  For patients with a device: patients will be at rest and the adjustments of their device will be made by a study physician or device coordinator, done routinely in clinical practice. This will take up to 15 minutes and during this time; participants will wear a face mask and breathing parameters are recorded using the SHAPE-HF system (SHAPE Medical St. Paul, MN) that measures respiratory airflow and the constituent respiratory gases, oxygen and carbon dioxide.
  Other Names: HeartMate 2; HeartWare; Biventricular pacemaker

SUMMARY:
To observe and document ventilation parameters in the advanced heart failure population, through the course of illness, which often includes cardiac resynchronization therapy (CRT), left ventricular assist device (LVAD), and transplant. Findings from this cohort are anticipated to be of sufficient interest to the scientific community to merit publication and are likely to provide preliminary data for future hypothesis generation and subsequent prospective, randomized controlled trials.

A compact, inexpensive apparatus has recently become commercially available for performing sub-maximal exercise testing (SHAPE Medical, St Paul, MN), including gas exchange analysis and will be used in this study. This apparatus is not investigational.

DETAILED DESCRIPTION:
Cardiopulmonary exercise testing (CPXT) has a long history in the evaluation and management of cardiovascular diseases, particularly in patients with advanced heart failure.

Cardiovascular exercise testing is a safe, well-developed, and validated method for risk stratification and objective documentation of exercise capacity in patients with severe heart failure (1,2). Recent studies have also shown that exercise testing has prognostic power for heart failure hospitalization and mortality (3,4), but limited published data are available in a large group of advanced heart failure patients, such as those with cardiac resynchronization therapy (CRT) and left ventricular assist devices (LVAD)

Advanced or suspected advanced heart failure. Typical patients screened for this study will be patients who have been referred to the University of Minnesota for evaluation for advanced heart failure options, such as cardiac transplant or mechanical circulatory support. This is a somewhat heterogeneous population, but all have been diagnosed by referring physician as having sufficiently severe heart failure to seek tertiary care. Most are anticipated to have severely depressed ejection fraction (<30% and typically <20%), but patients with preserved ejection fraction and either hypertrophy or restrictive cardiomyopathy will also be eligible. Patients pulmonary hypertension, on any therapy (other than diuretics alone), are also felt to be at high risk of developing right heart failure and may also be included. Patients who have already undergone LVAD or cardiac transplant are also considered to have advanced heart failure and are eligible to participate, regardless of the severity of their symptoms at the time of enrollment.

Healthy volunteers may be included for comparison.

This is a non-randomized, observational investigation of sub-maximal exercise ventilation parameters in patient diagnosed with, or suspected to have, advanced heart failure.

Duration of follow-up will be up to five years. Some subjects will undergo only one exercise test. Patients who present with heart failure but subsequently undergo CRT implantation, LVAD implantation, or cardiac transplant will be asked to repeat the submaximal exercise test. The timing between any of these events is unpredictable, so the duration of follow-up cannot be predicted. Subjects will be followed for change of status for up to 5 years. The total number of tests that any one person could potentially have is 5 (baseline plus one after each therapy), although we expect that most participants would not be asked to undergo more than 3 tests.

For patients without a device: Patients start at rest for 2 minutes and will wear a face mask and breathing parameters are recorded using the SHAPE-HF system (SHAPE Medical St. Paul, MN) that measures respiratory airflow and the constituent respiratory gases, oxygen and carbon dioxide. The SHAPE-HF system will continue to monitor and the patient then will start walking on a treadmill with a variable speed of 1-3 mph and a variable grade of 0-6%. The total treadmill time will be no more than 10 minutes.

For patients with a device: patients will be at rest and the adjustments of their device will be made by a study physician or device coordinator, done routinely in clinical practice. This will take up to 15 minutes and during this time; participants will wear a face mask and breathing parameters are recorded using the SHAPE-HF system (SHAPE Medical St. Paul, MN) that measures respiratory airflow and the constituent respiratory gases, oxygen and carbon dioxide. Device parameters will be returned to baseline settings following this part of the test.

Sub-maximal exercise testing approximately 30 minutes in duration will be performed on a treadmill at a slow and constant pace, the speed of the treadmill will range from 1-2 mph and the grade will range from 0-2% depending on the patient's exercise tolerance. The exercise will be split into two rounds of exercise up to 15 minutes each. Subjects may rest as long as they would like between the two tests.

The first round, participants will wear a face mask and breathing parameters are recorded using the SHAPE-HF system. (See section 13B for sample report).

In the second round, every two minutes, up to 15 minutes, participants will be asked to take 8 breaths using a breathing bag containing a standard mixture of gases (0.7% acetylene, 21% oxygen, 9% Helium and the balance of nitrogen)-this gas mixture is routinely used in pulmonary function laboratories to measure lung function and has the same amount of oxygen as room air. Acetylene mass spectroscopy is then used to measure cardiac output noninvasively.

Neither the SHAPE-HF system, nor the methods of gas exchange during exercise are investigational.

Participants who are treated with cardiac resynchronization therapy and/or ventricular assist device may have minor adjustments made to their device parameters every 2 minutes during the testing. The adjustments will be made by a study physician or device coordinator, as mentioned before, done in routine practice. Device parameters will be returned to baseline settings following the test.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Advanced heart failure suspected or diagnosed

Exclusion Criteria:

1. Inability to ambulate at least one block
2. Angina that has developed or a changed in pattern/symptoms since last physician visit.
3. Recent life-threatening arrhythmia or diagnosis that suggests high-risk of exacerbation of arrhythmia with exercise (catecholaminergic polymorphic ventricular tachycardia, e.g.)
4. LVAD driveline infection or suspected driveline infection
5. Medical activity restriction that precludes ambulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with, or suspected to have, advanced heart failure and who meet inclusion and exclusion criteria are eligible for participation. Those who have undergone LVAD implantation, heart transplantation or are on the transplant list, and those with biventricular pacemaker who meet study criteria are also eligible for study participation. Patients diagnosed with pulmonary hypertension and therefore at risk for developing right sided heart failure may also be included.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Sub-maximal exercise ventilation parameters | Pre and Post-LVAD placement
  Observational investigation of sub-maximal exercise ventilation parameters in patient diagnosed with, or suspected to have, advanced heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Eckman, MD, Principal Investigator — University of Minnesota
Locations (1):
- Masonic Clinical Research Unit, Minneapolis, Minnesota, United States